CLINICAL TRIAL: NCT05583669
Title: A Phase 1, Subject- and Investigator-Blinded, Sponsor-Unblinded, Placebo-Controlled, Randomized, Sequential Cohort Study to Assess the Safety and Pharmacokinetics of Multiple Ascending Subcutaneous Doses of DS-2325a in Healthy Subjects
Brief Title: A Study to Assess the Safety and Pharmacokinetics of Multiple Ascending Subcutaneous Doses of DS-2325a in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS2325-106
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Netherton Syndrome
Keywords: Netherton Syndrome; DS-2325a; Healthy Participants
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DS-2325a SC (Experimental): Participants who will be randomized to receive DS-2325a as a fixed dose subcutaneous (SC) injection (starting dose 300 mg).
  Interventions: Drug: DS-2325a
- Placebo SC (Experimental): Participants who will be randomized to receive placebo as a subcutaneous (SC) injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS-2325a — Subcutaneous injection (starting dose 300 mg)
  Arms: DS-2325a SC
Drug: Placebo — Subcutaneous injection
  Arms: Placebo SC

SUMMARY:
Netherton syndrome (NS) is a rare autosomal recessive disease and no systemic treatment or standard of care currently exists for patients with NS. DS-2325a, a specific and potent inhibitor of kallikrein 5, is expected to treat NS by replacing a defective gene.

DETAILED DESCRIPTION:
This study for DS-2325a will evaluate the safety, tolerability, and pharmacokinetics of multiple ascending doses of DS-2325a in healthy participants. DS-2325a will be evaluated after subcutaneous (SC) injections.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand a written informed consent, which must be obtained prior to initiation of study procedures.
* Must be willing and able to comply with all study requirements.
* Healthy males or non-pregnant, non-lactating healthy females.
* Aged 18 to 50 years of age (inclusive) at the time of signing informed consent.
* BMI of 18.0 kg/m^2 to 30.0 kg/m^2 (inclusive) as measured at Screening.
* Women of childbearing potential who are sexually active with a male partner must practice effective contraception during the study treatment period and for 90 days after last IMP administration. They must agree to use 2 different means of nonhormonal contraceptive methods.
* Women of non-childbearing potential must be either surgically sterile or in menopausal state confirmed as follows: 1 year of spontaneous amenorrhea without an alternative medical cause and a serum follicle stimulating hormone (FSH) level ≥40 mIU/mL.
* Male participants who are sexually active with a female partner of childbearing potential must use, with their partner, a condom plus an approved method of highly effective contraception from the time of informed consent until 90 days after last IMP administration.
* Women should not donate eggs and men should not donate sperm during the study treatment period and for at least 90 days after last IMP administration.
* All female participants must have a negative serum pregnancy test at Screening and Admission (Day -2).

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, metabolic, endocrine, immunologic, infectious, dermatologic, neurologic, oncologic, psychological, psychiatric, ophthalmologic, or gastrointestinal disease (except cholecystectomy), as judged by the Investigator.
* History or presence of chronic lung or respiratory disease, including clinically significant asthma (as judged by the Investigator) and chronic obstructive pulmonary disease (COPD).
* History, or presence in the average of triplicate ECGs at Screening and Admission (Day -2).
* Laboratory results (serum chemistry, hematology, coagulation, and urinalysis) outside the normal range, if considered clinically significant by the Investigator at Screening or Admission (Day -2).
* Creatinine clearance (CrCl) <80 mL/mina t Screening.
* History or presence of any other clinically significant condition, including laboratory abnormality, that in the opinion of the Investigator, would jeopardize the safety of the participant, obtaining informed consent, compliance to the study procedures, or the validity of the study results.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Any Treatment-emergent Adverse Events Following Administration of DS-2325a | Screening (Day -28 to -3) pre-dose up to Day 78 post-dose
  Treatment-emergent adverse events (TEAEs) are defined as new adverse events (AEs) that occur after the dose of study drug or as AEs that were present prior to the dose of study drug but which worsened in severity after the start of study drug.

SECONDARY OUTCOMES:
Pharmacokinetic Parameter Area Under the Concentration Curve (AUCtau) | Day 1: pre-dose & 4, 8, 24, 72, 96, 120, 144 hours (hr) post-dose; Day 8 & 14: pre-dose; Day 22: pre-dose & 4, 8, 24, 48, 72, 96, 120, 144, 168 hr post-dose; Day 36, 43, 57, & 78
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Maximum Concentration (Cmax) | Day 1: pre-dose & 4, 8, 24, 72, 96, 120, 144 hours (hr) post-dose; Day 8 & 14: pre-dose; Day 22: pre-dose & 4, 8, 24, 48, 72, 96, 120, 144, 168 hr post-dose; Day 36, 43, 57, & 78
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Average Concentration (Cavg) | Day 1: pre-dose & 4, 8, 24, 72, 96, 120, 144 hours (hr) post-dose; Day 8 & 14: pre-dose; Day 22: pre-dose & 4, 8, 24, 48, 72, 96, 120, 144, 168 hr post-dose; Day 36, 43, 57, & 78
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Drug Accumulation Ratio for AUCtau and Cmax (Rac) | Day 1: pre-dose & 4, 8, 24, 72, 96, 120, 144 hours (hr) post-dose; Day 8 & 14: pre-dose; Day 22: pre-dose & 4, 8, 24, 48, 72, 96, 120, 144, 168 hr post-dose; Day 36, 43, 57, & 78
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) | Day 1: pre-dose & 4, 8, 24, 72, 96, 120, 144 hours (hr) post-dose; Day 8 & 14: pre-dose; Day 22: pre-dose & 4, 8, 24, 48, 72, 96, 120, 144, 168 hr post-dose; Day 36, 43, 57, & 78
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Terminal Elimination Half-life (T1/2) | Day 1: pre-dose & 4, 8, 24, 72, 96, 120, 144 hours (hr) post-dose; Day 8 & 14: pre-dose; Day 22: pre-dose & 4, 8, 24, 48, 72, 96, 120, 144, 168 hr post-dose; Day 36, 43, 57, & 78
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Elimination Rate Constant Associated With the Terminal Phase (Kel) | Day 1: pre-dose & 4, 8, 24, 72, 96, 120, 144 hours (hr) post-dose; Day 8 & 14: pre-dose; Day 22: pre-dose & 4, 8, 24, 48, 72, 96, 120, 144, 168 hr post-dose; Day 36, 43, 57, & 78
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Number of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) | Day 1: pre-dose and Days 15, 22, 36, 57, and 78
  Blood samples will be collected to determine ADAs.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Daiichi Sankyo
Locations (1):
- Quotient Sciences -Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/